CLINICAL TRIAL: NCT06669793
Title: A Randomized Trial Comparing the Biolimus-coated Balloon and Paclitaxel-coated Balloon in de Novo Large Vessel Coronary Lesions
Brief Title: Biolimus-Coated Balloon in de Novo Large Vessel Coronary Lesions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Third People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-02-008-H01
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Coronary Arterial Disease (CAD)
Keywords: paclitaxel-coated balloon; biolimus-coated balloon; de novo lesions; large coronary artery vessel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biolimus-coated balloon group (Experimental)
  Interventions: Device: biolimus-coated balloon
- paclitaxel-coated balloon group (Experimental)
  Interventions: Device: paclitaxel-coated balloon

INTERVENTIONS:
Device: biolimus-coated balloon — 238 subjects with de novo large vessel coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of Biolimus-coated balloon.
  Other Names: BA9 balloon
  Arms: biolimus-coated balloon group
Device: paclitaxel-coated balloon — 237 subjects with de novo large vessel coronary lesions who met the inclusion/exclusion criteria were enrolled; subjects were assigned to the treatment group of paclitaxel-coated balloon.
  Arms: paclitaxel-coated balloon group

SUMMARY:
Percutaneous coronary intervention (PCI) is one of the standard treatments for patients with acute and chronic coronary syndromes that are consistently recommended by current national and international guidelines. Currently, even with the most advanced design concepts of drug-eluting stents (DES), the permanent foreign body and in-stent restenosis after implantation are still very detrimental to the clinical outcomes of patients. These problems have been mitigated to some extent by the advent of the drug-coated balloon (DCB), a special balloon coated with an antiproliferative drug that is uniformly delivered to the vessel wall during endovascular dilatation to inhibit endothelial proliferation.

This study is a prospective randomized study of a novel drug-coated balloon for the treatment of de novo coronary artery large vessel lesions. By comparing the clinical outcomes of the novel BA9 drug-coated balloon (BCB) with those of the paclitaxel-coated balloon (PCB) in the treatment of de novo coronary artery large vessel, we evaluated the safety and efficacy of the BCB for such lesions, and provided evidence for the later use of rapamycin-based drug-coated balloons in PCI.

They are randomly dividing them into BCB treatment group and PCB treatment group according to the ratio of 1:1. All subjects accept clinical follow-up after operation, at 30 days, 6 months, 9 months and 12 months after operation.

ELIGIBILITY:
Inclusion Criteria:

* Radiography inclusion criteria

  1. angiographically confirmed de novo coronary artery lesion;
  2. target lesion stenosis must be ≥70% or ≥50% with clear evidence of myocardial ischaemia (visual assessment);
  3. target lesion vessel diameter is between 2.75mm and 4.0mm, target lesion length must be ≤25mm (visual assessment);
  4. either one or two target lesions to be treated; if two target lesions, they must be located in different target vessels;
  5. successful target lesion preparation: residual stenosis ≤30%, no flow-restricting entrapment, and TIMI grade 3 flow; General inclusion criteria

  <!-- -->

  1. subjects at the age between ≥18 and ≤80 years old;
  2. patients with symptoms or evidence of myocardial ischaemia;
  3. subjects are willing to participate in the study, sign informed consent form, and accept clinical follow-up after operation and at 30 days, 6 months, 9 months and 12 months after operation.

Exclusion Criteria:

* Radiography exclusion criteria

  1. in-stent lesions;
  2. For the left main disease, true bifurcation lesion, chronic total occlusive lesions;
  3. Severely calcified lesions and tortuous lesions; lesions that have failed pretreatment; lesions unsuitable for balloon delivery and dilatation;
  4. Previous use of any brand of drug-coated balloon in the target vessel. General inclusion criteria

  <!-- -->

  1. Any patient with myocardial infarction within one month;
  2. Patients with severe congestive heart failure (NYHA Level IV severe heart failure) or severe valvular heart disease; or left ventricular ejection fraction of less than 35%;
  3. Patients with stroke, peptic ulcer or gastrointestinal bleeding within the past 6 months; or patients with bleeding tendency or coagulation disorders;
  4. Patients with severe liver failure (ALT and AST are larger than 3 times of the upper limit of normal value), who are judged to be not applicable to angiography by investigators;
  5. Patients with severe renal failure(eGFR<30ml/minute) or such medical history, failure to comply with angiography conditions;
  6. Subjects who are intolerance or allergic to heparin, contrast agent, Biolimus, polyethylene oxide and polylactic acid - glycolic acid polymer;
  7. Patients who plans to accept selective operation within 1 year;
  8. Patients who are participating in the clinical trial of other drug or device without reaching the time limit of primary endpoint;
  9. Subjects who are considered to be not applicable to be enrolled by investigators due to other reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 475 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2027-05-23 (Estimated); Study Completion 2028-05-23 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 12 months
  include cardiac death, non-fatal myocardial infarction, and target lesion revascularization.

IPD SHARING:
Plan to Share IPD: Undecided